CLINICAL TRIAL: NCT05339074
Title: Maintenance Ketamine Infusions for Treatment-Resistant Bipolar Depression: An Open-Label Extension Trial
Brief Title: Maintenance Ketamine Infusions for Treatment-Resistant Bipolar Depression
Acronym: KET-BD-Sustain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua Rosenblat (Other)
Responsible Party: Sponsor-Investigator, Joshua Rosenblat, Principal Investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-5963
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental): Open-label ketamine infusions will be provided on a flexible schedule (every 2-4 weeks) with flexible dosing (0.5-1.0mg/kg over 40 minutes) titrated to optimize benefits, while minimizing the dosage and frequency over a 12-week extension period
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — 60 patients will receive ketamine hydrochloride over 12 weeks, flexible dosed between 0.5 mg/kg to 1.0 mg/kg

SUMMARY:
Growing evidence has supported rapid and robust antidepressant effects with subanesthetic doses of intravenous (IV) ketamine for treatment resistant depression (TRD). However, no completed or ongoing RCTs have evaluated the effects of repeated doses of IV ketamine for a homogenous sample of patients with treatment-resistant bipolar disorder depression (TRBD). The primary research goal is to determine the acute antidepressant efficacy, safety and tolerability of repeated sub-anesthetic maintenance doses of IV ketamine in, over a period of twelve weeks. Open-label ketamine infusions will be provided on a flexible schedule (every 2-4 weeks) with flexible dosing (0.5-1.0mg/kg over 40 minutes) titrated to optimize benefits, while minimizing the dosage and frequency over a 12-week extension period. All patients participating in this open-label study will have completed an acute course of infusions in a parent two-site, phase II, double-blinded midazolam-controlled RCT trial. In addition to this acute course of four infusions, a maximum of six infusions will be provided over the 12-week period. Secondary aims include evaluating effects of IV ketamine on suicidal ideations, quality of life, function and duration of effects. Herein, a two-site (University Health Network and Ontario Shores Centre for Mental Health Sciences), single-arm, open label, 12-week extension trial evaluating the effects of flexibly-dosed adjunctive ketamine infusions for TRBD to maintain antidepressant effects in participants who achieved an antidepressant response (MADRS decrease by >50%) or remission (MADRS < 12) following an acute course of four ketamine infusions is proposed. The primary outcome will be Montgomery-Åsberg Depression Rating Scale (MADRS) scores, determining by a linear mixed model from baseline to week 12. Secondary outcomes include evaluating response and remission rates, safety, tolerability (including treatment-emergent mania), and effects on suicidality, anxiety, quality of life, function and the duration of effects.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, voluntary informed consent prior to study enrollment. Substitute decision makers will not be allowed to consent to study on a potential patient's behalf.
2. Male or female between the age of 21 to 65, inclusive.
3. Meets DSM-5 criteria for Bipolar I or II Disorder, currently experiencing a Major Depressive Episode without psychotic features. Diagnosis confirmed by study psychiatrist at the start of the parent KET-BD randomized clinical trial (RCT).
4. Patients in the KET-BD RCT 4a. Patients in the ketamine arm of the KET-BD RCT must have experienced an antidepressant response (i.e. change in MADRS score ≥ 50% at day 14 compared to baseline or Clinical Global Impression-Improvement (CGI-I) = 2 'much improved' or 1 'very much improved') or experienced clinical remission of symptoms (i.e., MADRS score < 12 on day 14) 4b. Patients in the midazolam arm of the KET-BD RCT must present as moderately to severely depressed (MADRS >21) on days 14 and 28 of the parent RCT and must be responders or remitters following four flexibly dosed infusions over 2 weeks.
5. Current depressive episode has inadequate response to two or more adequate first-line treatment trials for bipolar depression, as per the 2018 CANMAT Bipolar Disorder Guidelines. First line treatment trials include the use of lithium, valproate, carbamazepine, lamotrigine and/or any antipsychotic medication. Adequate medications confirmed at the start of the parent KET-BD RCT.
6. Patient must be receiving guideline-concordant pharmacotherapy without changes in the last month, including a therapeutic dose of a mood stabilizer.

Exclusion Criteria:

1. Currently exhibiting symptoms of mania, hypomania, or mixed state bipolar, as determined by the Young Mania Rating Scale (YMRS) score greater than 12.
2. Current symptoms of psychosis or a substance use disorder within the past 3 months. History of psychotic features during a mood episode will not be excluded.
3. History of neurological disorders (including, but not limited to, uncontrolled seizure disorder, history of stroke within past 12 months, major head injuries, aneurysmal vascular disease [including thoracic and abdominal aorta, intracranial, and peripheral arterial vessels], arteriovenous malformation, or intracerebral hemorrhage)
4. Lifetime history of a primary psychotic disorder (including, but not limited to, schizophrenia or schizoaffective disorder)
5. Lifetime history of ketamine use disorder
6. Presence of active suicidality, requiring involuntary inpatient treatment or recent suicide attempts within the past 3 months.
7. Presence of a contraindication to ketamine, including a drug allergy, uncontrolled hypertension (baseline systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg), low or labile blood pressure, myocardial infarction within past 12 months, cardiac arrhythmia, moderate to severe hepatic impairment (i.e., Child-Pugh score of B or C), moderate or severe renal impairment (glomerular filtration rate (GFR) < 45 milliliters/min), heart failure, or coronary artery disease
8. Pregnant or breastfeeding women or women who intend to get pregnant. Patients who are sexually active must agree to use a highly effective contraceptive method (as outlined in section 5.9).
9. Use of prohibited concomitant medications, including other forms of ketamine or esketamine, benzodiazepines, monoamine oxidase inhibitors, stimulants, medical or recreational cannabis of any form.
10. Patients in the ketamine-arm of the parent RCT, that did not reasonably tolerate 4 infusions of flexibly-dosed ketamine, as determined by the investigator and/or patient

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in depression severity using the Montgomery-Asberg Depression Rating Scale (MADRS) | 12 weeks
  The MADRS is a clinician-rated scale measuring depression severity. It consists of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60. A higher score is indicative of greater depressive severity. Response rates are defined as > 50% decrease and Remission <12 actual score.

SECONDARY OUTCOMES:
Recruitment and Retention Rates | 12 weeks
  The feasibility of ketamine as a treatment in bipolar disorder will be measured by recruitment and retention rates.
Treatment-Emergent Adverse Events | 12 weeks
  Treatment-emergent adverse events will be assessed using patient-reported adverse events.
Suicidality | 12 weeks
  Suicidality will be assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS) which is a clinical assessment used to assess suicidal ideation and suicidal behaviour. It measures the incidence of suicidality via "yes" or "no" questions as well as the severity of suicidal ideation if present on a scale of 1 to 5 with 5 being the most severe.
Treatment-Emergent Mania | 12 weeks
  Treatment-emergent mania will be assessed using the Young Mania Rating Scale (YMRS) which is a clinical assessment used to evaluate manic symptoms and their severity. It consists of 11 items with a maximum possible score of 60, with higher scores indicating more severe manic symptoms.
Quality of Life (QOL) | 12 weeks
  Quality of life will be assessed using the Quality of Life-BD (QOL.BD) scale, which contains 56 questions over 12 domains. It uses a 5-component scale that evaluates mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This scale is numbered from 56 to 280, 280 indicating a high quality of life, while 56 denotes a low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rosenblat, MD, MSc, Principal Investigator — Toronto Western Hospital, Psychiatry
Locations (3):
- Canada (3):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: No